CLINICAL TRIAL: NCT02546453
Title: Use of Specific Genetic Alteration s of Tumoral Cells Identified by NGS to Follow Peripheral Samples of Children With Metastatic and/or High Risk Solid Tumor -
Brief Title: Use of Specific Genetic Alteration s of Tumoral Cells Identified by the Next Generation Sequencing Techniques (NGS) to Follow Peripheral Samples of Children With Metastatic and/or High Risk Solid Tumor - NGSKids
Acronym: NGSKids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2014-01
Record Dates: First submitted 2015-04-23; First posted 2015-09-10 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Metastatic and/or High Risk Solid Tumor of Children
Keywords: high risk solid tumor pediatric, genetic alteration, Metastatic solid tumor pediatric
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumoral specific genetic alterations (Other): NGS techniques (next generation sequencing) will be used to identify specific genetic alterations of tumoral cells of a patient. If specific genetic alterations is detected, they will be used to detect circulating tumor DNA and/or circulating/disseminated tumoral cells (CTC/DTC) in peripheral samples (blood, bone marrow, cerebral spinal fluid) collected before, during and after treatment.
  Interventions: Biological: Tumoral specific genetic alterations

INTERVENTIONS:
Biological: Tumoral specific genetic alterations — A buccal swab and a blood sample will be used at the diagnostic to identify the specific genetic alterations of tumoral cells.
Biological: Tumoral specific genetic alterations — Collection of blood (maximum 9 samples of 3 to 5 ml), bone marrow (maximum 3 samples of 3 to 5 ml) and cerebral spinal fluid (maximum 3 samples 500µl to 1ml).

SUMMARY:
The search for genetic alterations in primary tumor by NGS techniques followed by the detection of these alterations in circulating tumor DNA and/or CTC/DTC present in peripheral samples (blood, cerebrospinal fluid, bone marrow, possibly urine) collected during several steps and after the treatment could be a tool to monitor the response during and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with metastatic and/or high risk solid tumor, of the following pathologies :

Neuroblastoma, sarcoma, malignant brain tumor (medulloblastoma, high-grade glioma), bone tumors, rhabdoid tumors, others rare tumors

* Availability of a frozen tumoral sample (primary tumor or metastasis whatever the localization) at diagnosis allowing analysis of genetic alterations by a NGS technique
* Age < 18 years
* Signed informed consent by parents or legal representatives
* Patient having health care insurance

Exclusion Criteria :

* Age ≥ 18 years
* No signed informed consent by parents or legal representatives

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Detection by Polymerase Chain Reaction (PCR) of specific genetic alterations | at the inclusion
  Genetic alterations which have been previously detected by NGS technique in the tumor, in circulating tumoral DNA and/or CTC/DTC present in a blood sample at the inclusion.
Detection of specific genetic alterations of tumoral cells in peripheral samples | Up to 6 years
  Detection of specific genetic alterations of tumoral cells in peripheral samples for which presence of tumoral cells has been confirmed by conventional clinic techniques (cytology, anatomopathology, immunohistochemistry

SECONDARY OUTCOMES:
Detection of genetic alterations in solid tumor pediatric samples | At the inclusion
  Use of identified genetic alterations in solid tumor pediatric samples to help to confirm diagnosis and prognosis and to search for new therapeutic targets
Change of CTC/DTC/circulating tumoral DNA levels detected by PCR targeting specific genetic alterations of tumoral cells in peripheral samples will be confronted to clinical features including patient outcome | Up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).